CLINICAL TRIAL: NCT05755334
Title: Ropivacaine Pharmacokinetics After Erector Spinae Block in Children Undergoing Posterior Spinal Fusion
Brief Title: Ropivacaine Pharmacokinetics After Erector Spinae Block
Acronym: PK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gianluca Bertolizio, Principle Inverstigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-9498
Record Dates: First submitted 2023-02-10; First posted 2023-03-06 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pain; Spinal Fusion
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, single blinded, randomized non-superiority study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine 0.1% (Active Comparator): Erector spinae plane block with 2 ml/kg of ropivacaine 0.1%.
  Interventions: Drug: Ropivacaine
- Ropivacaine 0.2% (Experimental): Erector spinae plane block with 1 ml/kg of ropivacaine 0.2%.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Administration of Ropivacaine

SUMMARY:
The primary aim is to evaluate the analgesic efficacy of either technique by measuring cumulative morphine consumption in the first 24 hours after an erector spinae plane block with 2 ml/kg of ropivacaine 0.1% (2 ml/kg) or 1 ml/kg of ropivacaine 0.2%.

The secondary aim of this study is to describe the pharmacokinetics of ropivacaine 0.1% and ropivacaine 0.2% after erector spinae block in children undergoing posterior spinal fusion.

DETAILED DESCRIPTION:
Pain is of particular concern in pediatric patients undergoing posterior spinal fusion surgery. In children, posterior spinal fusion is performed for neuromuscular or adolescent idiopathic scoliosis. Posterior spinal fusion is highly invasive and entails the fusion of multiple adjacent vertebral bodies. The surgery generates profound pain from multiple tissue sources including bones, ligaments, intervertebral discs, nerve root sleeves, fascia and muscles. In these patients, greater perioperative pain has been shown to increase the risk of chronicity, prolonged pain medication use, delayed rehabilitation and delayed return of function. Patients experiencing moderate-to-severe pain in the acute postoperative period were more likely to report higher levels of pain severity, use more pain medication, and miss a greater number of school/workdays due to back pain in the last three month.

The mainstream perioperative pain therapy in patients undergoing posterior spinal fusion is opioid-based. Prolonged intravenous opioids, however, are associate to prolonged length of stay. As a results, adjuvants of such as acetaminophen, nonsteroidal anti-inflammatory drugs and ketamine are routinely used in some centers.

Recently, the erector spinae plane (ESP) block has been proposed as an effective adjuvant in the multimodal analgesia after posterior spinal fusion .

The erector spinae plane block is a paraspinal fascial plane block in which the needle placement is between the erector spinae muscle and the thoracic transverse processes, and a local anesthetic is administered, blocking the dorsal and ventral rami of the thoracic and abdominal spinal nerves. This blockage of the dorsal and ventral rami of the spinal nerves helps to achieve a multi-dermatomal sensory block of the anterior, posterior, and lateral thoracic and abdominal walls. The erector spinae plane block has been successfully implemented in the multimodal analgesia management in both adults and children.

However, there is limited information about the pharmacokinetics of ropivacaine after erector spinae plane blocks. In adults, studies reported potentially neurotoxic plasma concentrations after the injection of a 'safe" (100 mg) dose of ropivacaine in the transversus plane. In contrast, in children, plasma concentrations of ropivacaine after ilioinguinal-iliohypogastric, transversus plane block appear to remain well below the neurotoxic blood concentration for total ropivacaine (2.2 μg/ml). Similarly, plasma concentration after erector spinae plane block have been reported to be safe, but data are limited to a single small investigation. A recent pilot study in children showed high blood concentrations (0.56 μg/L) of unbound ropivacaine exceeding its potential neurotoxic blood concentration (0.15 μg/L), but concentrations of total ropivacaine below the neurotoxic (and cardiovascular) threshold. after erector spinae plane block with ropivacaine at high concentrations (0.5%).

In 2021, at the Montreal Children's Hospital (MCH) an Enhanced recovery after surgery (ERAS) protocol for patients undergoing posterior spinal fusion was implemented. This protocol includes standardized intraoperative anesthesia and postoperative analgesia (Annex 1). At the end of the surgery, after confirming adequate spinal cord function with the motor and somatosensory evoked potentials and before skin closure, surgeon injects a 2 mg/kg dose of the local anesthetic ropivacaine 0.1% (total volume 2 ml/kg) or 0.2% (total volume 1 ml/kg) in the erector spinae plane.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 8 year older and > 25 kg undergoing posterior spinal fusion surgery
* Parents or legal guardians that are fluent in French of English

Exclusion Criteria:

* Patients with any contraindication to locoregional anesthesia
* Patients that are expected to be intubation for a prolonged period of time after surgery
* Patients with anemia (hematocrit < 30%) before surgery or at time of the first study blood draw
* Patients that do not receive an erector spinae plane block
* Parents or legal Patient/legal guardian that to not consent to participate in the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | 24 hours after surgery
  Total opioid consumption after surgery
Pain after surgery | 24 hours after the surgery
  Severity of pain after surgery measured by heart rate variability
Pain during surgery | During the the surgery
  Severity of pain during surgery during measured by heart rate variability
Post-operative Complications | 24 hours after the surgery
  The number of anesthesia and surgical related complications

SECONDARY OUTCOMES:
Secondary outcome | During the and 24 hours after the surgery
  The secondary outcome of this study is defined as the difference in rate in which of ropivacaine 0.1% and ropivacaine 0.2% is absorbed after a spinal block in children undergoing posterior spinal fusion

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engelhardt, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre